CLINICAL TRIAL: NCT01797146
Title: Effectiveness of Catheter Reminder and Evaluation (CARE) Program in Reducing the Catheter-day and Prevention of Catheter-associated Infections
Brief Title: Effectiveness of Catheter Reminder and Evaluation Program
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Pinyo Rattanaumpawan, Assistant Professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 656/2555(EC1)
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: All Hospitalized Patients; With and Without Catheter
MeSH Terms: interventions — Program Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARE (Active Comparator): All patients in the intervention wards will receive the Catheter Reminder and Evaluation (CARE) intervention.
  Interventions: Procedure: Catheter Reminder and Evaluation Program
- Control (No Intervention): All patients in the control wards will receive usual care without the CARE intervention.

INTERVENTIONS:
Procedure: Catheter Reminder and Evaluation Program — This intervention will be implemented by ward nurses and responsible physicians. The details of intervention are shown below.
  1. Nurse: Every morning, a ward nurse will check if any patient has a urinary catheter or a central venous catheter in place. An order sheet will be marked with a CARE-rubber stamp and the following information will be added by hand-writing.
     * Type and duration of urinary catheter use.
     * Indication of urinary catheter _________
     * Type and duration of central venous catheter use
     * Indication of urinary catheter _________
  2. Responsible physician: During a morning round, a physician needs to fill the indication of catheter use. If a given physician does not fill the indication of urinary catheter use, the catheter will be automatically removed. If a given physician does not fill the indication of central venous catheter, the CARE team will be notified.
  Arms: CARE

SUMMARY:
The investigators will conduct a cluster randomized controlled trial to evaluate the efficacy of Catheter Reminder and Evaluation program (CARE) in reducing the duration of catheter use and the number of infection relating to catheter use.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized adults in 6 general medical wards at Siriraj Hospital
* With or Without catheter

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Urinary catheter day | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Total duration of urinary catheter use (day)

SECONDARY OUTCOMES:
CA-UTI | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Number of catheter-associated urinary tract infection episode

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand